CLINICAL TRIAL: NCT07124468
Title: A Phase 1, Randomized, Open-Label, Trial Evaluating the Plasma, Epithelial Lining Fluid, and Alveolar Macrophage Concentrations of Intravenous Meropenem-Pralubactam(Meropenem/FL058) in China Healthy Adult Participants
Brief Title: Assess the Plasma, Epithelial Lining, and Alveolar Macrophage Concentrations of Intravenous Meropenem-Pralubactam (Meropenem/FL058) in China Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FL058-Ⅰ-05
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intravenous Meropenem-Pralubactam (Experimental)
  Interventions: Drug: Meropenem-Pralubactam

INTERVENTIONS:
Drug: Meropenem-Pralubactam — The study is designed to enroll approximately 16 healthy participants. The study will evaluate the plasma, epithelial lining fluid, and alveolar macrophage concentrations of Meropenem-Pralubactam

SUMMARY:
The goal of this clinical trial is to evaluate the Epithelial Lining Fluid concentrations and permeability of Intravenous Meropenem-Pralubactam(Meropenem/FL058) in China Healthy Adult Participants. The main question it aims to answer is:

• [question 1] : What are the concentrations of meropenem and Pralubactam in plasma, epithelial lining fluid (ELF), and alveolar macrophages (AM) at each time point

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-45 years
* Body mass index (BMI): 19-28 kg/m² , with body weight ≥50 kg.
* Pulmonary function at screening:

  1. Forced expiratory volume in 1 second (FEV₁) measured/predicted >80%
  2. Forced vital capacity (FVC) measured/predicted >80%
  3. All other ventilation and diffusion parameters normal or with no clinical significance.
* Participant capability:

  1. Ability to communicate effectively with investigators
  2. Willingness to comply with study procedures
  3. Voluntary participation with acceptance of bronchoalveolar lavage (BAL)
  4. Provision of written informed consent.
* Reproductive planning:

  1. No pregnancy, sperm/egg donation plans from signing informed consent through 28 days after last dose
  2. Participant and partner must use protocol-approved contraception.

Exclusion Criteria:

* Hypersensitivity to cephalosporins or carbapenem antibiotics.
* History or current diagnosis of respiratory system diseases.
* History or current diagnosis of coagulation disorders.
* Clinically significant diseases in cardiovascular, endocrine, neurological, digestive, hematological, metabolic, or psychiatric systems judged by the investigator to interfere with study outcomes.
* History of smoking or positive nicotine test during screening.
* Prior surgery involving pharynx, trachea/bronchi, or lungs.
* Drug abuse history within 1 year prior to screening or positive urine drug screen at screening.
* Alcohol intake >14 units/week on average within 6 months prior to screening.
* Participation in other clinical trials with investigational drugs/devices within 3 months prior to screening.
* Blood donation/loss ≥400 mL or blood product transfusion within 3 months prior to screening.
* Respiratory infections (bacterial/fungal/viral) within 2 weeks prior to screening (e.g., upper/lower respiratory tract infections).
* Use of any medication/vaccination within 14 days prior to screening or planned vaccination during the study.
* Clinically significant abnormalities in physical examination, 12-lead ECG, or imaging at screening per investigator's judgment.
* Pregnancy, lactation, or positive serum pregnancy test at screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-09-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
CPlasma、CELF、CAM | 5 days
  Assessment of plasma, ELF and AM concentrations of Intravenous Meropenem-Pralubactam after 4 doses of Meropenem-Pralubactam

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, China